CLINICAL TRIAL: NCT06209021
Title: Effects of Hyperbaric Oxygen Therapy on Middle and Inner Ear Functions
Acronym: HBOT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nahla Ahmed Abd elhafez Mousa, Principle investigator, Assiut University
Other Study IDs: Audiology2024
Record Dates: First submitted 2024-01-04; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Middle Ear Barotrauma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The goal of this observational study is to measure the effect of hyperbaric oxygen therapy on middle ear pressure in order to predict the risk factors for middle ear barotrauma also, to assess its effects on hearing functions of the inner ear in participant population. The main questions aim to answer are:

* Is there a change in middle ear pressure before and after exposure to hyperbaric oxygen therapy ?
* Is there a change in hearing threshold level before and after exposure to hyperbaric oxygen therapy ? The middle ear pressure, eustachian tube functions and the hearing threshold of the participants will be assessed immediately before the fist session and within one hour after the first and tenth sessions.

DETAILED DESCRIPTION:
Fifty four patients already treated by hyperbaric oxygen therapy recruited from hyperbaric oxygen therapy center of Assiut university hospitals. Otoscopic examination for all patients must be done before and after the session , assessment of middle ear pressure and the state of the eustachian tube through doing eustachian tube function tests (Valsalva and Toynbee tests for ears with intact tympanic membrane and modified inflation - deflation tests for ears with perforated tympanic membrane) by tympanometry for all patients before and after the first session of hjyperbaric oxygen therapy and after completion of the tenth session. Assessment of the hearing threshold level of the patients immediately before the first session and after the tenth session of hyperbaric oxygen therapy through doing pure tone audiometry ( air conduction and bone conduction audiometry) and speech audiometry to assess the speech discrimination score for the patients

ELIGIBILITY:
Inclusion Criteria:

* Patients of at least 18 years old.
* Patients accept participation in the research.
* Patients with out history of middle ear diseases.

Exclusion Criteria:

* Patients under age of 18 years old.
* Patients have middle ear effusion.
* Patients refuse to participate in the research.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients of both sexes already recommended to be treated by hyperbaric oxygen therapy for various medical conditions in hyperbaric oxygen therapy center.
Sampling Method: Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Measuring the changes of the middle ear pressure after exposure to hyperbaric oxygen therapy | Immediately before exposure to the first session of hyperbaric oxygen therapy and within one hour after exposure to the first and tenth session of hyperbaric oxygen therapy.
  Tympanometric assessment of the middle ear pressure and eustachian tube functions